CLINICAL TRIAL: NCT01460160
Title: A Phase 2 Multi-Center, Historically Controlled Study of Dasatinib Added to Standard Chemotherapy in Pediatric Patients With Newly Diagnosed Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Brief Title: Pediatric Philadelphia Positive Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Children's Oncology Group (Network); EsPhALL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-372; 2011-001123-20 (EudraCT Number); AALL1122 (Other: COG)
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Leukemia, Pediatric
MeSH Terms: conditions — Leukemia | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Dasatinib (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 60 mg/m2, Once daily, 2 years or until unacceptable toxicity
  Other Names: Sprycel

SUMMARY:
The purpose of this study is to determine whether Dasatinib when added to standard chemotherapy is effective and safe in the treatment of pediatric philadelphia chromosome positive acute lymphoblastic leukemia

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Newly diagnosed Philadelphia chromosome positive Acute Lymphoblastic Leukemia (ALL)
* Age >1 year and < less than 18 years old
* Induction chemotherapy ≤ 14 days according to institutional standard of care
* Adequate liver, renal and cardiac function

Exclusion Criteria:

* Prior treatment with a Oncogene fusion protein (BCR-ABL) inhibitor
* Extramedullary involvement of the testicles
* Active systemic bacterial, fungal or viral infection
* Down syndrome

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2012-04-13 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (127):
- United States (88):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Phoenix Children'S Hospital/Ctr. For Cancer & Blood Ctr., Phoenix, Arizona
  - University Of Arkansas For Medical Sciences, Little Rock, Arkansas
  - Antranik Agop Bedros, Loma Linda, California
  - Miller Children's and Women Hospital, Long Beach, California
  - Children'S Hospital Of L.A., Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Lpch & Sumc, Palo Alto, California
  - Kaiser Medical Center, Roseville, California
  - Ucsf - Hematology/Oncology, San Francisco, California
  - Children'S Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - A. I. Dupont Hospital For Children, Wilmington, Delaware
  - Children'S National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - University Of Florida, Gainesville, Florida
  - Nemours Children'S Clinic, Jacksonville, Florida
  - Md Anderson Cancer Center Orlando, Orlando, Florida
  - Nemours Childrens Hospital, Orlando, Florida
  - All Children'S Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - St. Mary'S, West Palm Beach, Florida
  - Children's Healthcare Of Atlanta, Atlanta, Georgia
  - Kapiolani Medical Center For Women & Children, Honolulu, Hawaii
  - Mountain States Tumor Institute, Boise, Idaho
  - Ann & Robert H Lurie Children's Hospital Of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Southern Illinois University School Of Medicine, Springfield, Illinois
  - James Whitcomb Riley Hospital For Children, Indianapolis, Indiana
  - Children'S Center For Cancer And Blood Diseases, Indianapolis, Indiana
  - University Of Kentucky, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Children'S Hospital Of Michigan, Detroit, Michigan
  - Helen Devos Children'S Hospital, Grand Rapids, Michigan
  - Michigan State University, Lansing, Michigan
  - Childrens Hospitals And Clinics Of Minnesota, Minneapolis, Minnesota
  - Univ Of Mississippi Med Ctr, Jackson, Mississippi
  - University Of Missouri Health Care, Columbia, Missouri
  - Children'S Mercy Hospital And Clinics, Kansas City, Missouri
  - Washington University Medical Center, St Louis, Missouri
  - Children'S Specialty Center Of Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Goryeb Children'S Hospital, Morristown, New Jersey
  - The Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - University Of New Mexico, Albuquerque, New Mexico
  - New York University, New York, New York
  - The Herbert Irving Pavilion, New York, New York
  - New York Presbyterian/Weill Cornell, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children'S Hospital, Columbus, Ohio
  - The Children'S Medical Center Of Dayton, Dayton, Ohio
  - The Toledo Children'S Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital & Health Center, Portland, Oregon
  - Oregon Health & Sci Univ, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children'S Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital Of Pittsburgh Of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - East Tennessee Children'S Hosp, Knoxville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Dell Children'S Medical Center Of Central Texas, Austin, Texas
  - Driscoll Children'S Hospital, Corpus Christi, Texas
  - Ut Southwestern, Dallas, Texas
  - Cook Children'S Hem/Onc Center, Fort Worth, Texas
  - Texas Children'S Cancer Center, Houston, Texas
  - Scott & White - McLane Children's Specialty Clinic, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Inova Pediatric Specialty Center Ii, Fairfax, Virginia
  - Children'S Hosp-Kings Daughter, Norfolk, Virginia
  - Seattle Children'S, Seattle, Washington
  - St Vincent Hospital, Green Bay, Wisconsin
  - Kenneth Desantes, Md, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Local Institution, Sth Brisbane, Queensland
  - Local Institution, Parkville, Victoria
  - Local Institution, Nedlands, Western Australia
- Canada (7):
  - Alberta Children'S Hospital, Calgary, Alberta
  - Stollery Children'S Hospital, Edmonton, Alberta
  - Local Institution, London, Ontario
  - Children'S Hospital Of Eastern Ontario, Ottawa, Ontario
  - Chu Ste-Justine, Montreal, Quebec
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Italy (11):
  - Local Institution, Bologna
  - Local Institution, Cagliari
  - Local Institution, Catania
  - Local Institution, Florence
  - Local Institution, Genova
  - Local Institution, Monza
  - Local Institution, Napoli
  - Local Institution, Palermo
  - Local Institution, Roma
  - Local Institution, Torino
  - Local Institution, Trieste
- Local Institution, San Juan, Puerto Rico
- United Kingdom (17):
  - Local Institution, Bristol, Avon
  - Local Institution, Cardiff, Glamorgan
  - Local Institution, Aberdeen, Grampian
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Southampton, Hampshire
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Edinburgh, Lothian
  - Local Institution, Liverpool, Merseyside
  - Local Institution, Leeds, North Yorkshire
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Oxford, Oxfordshire
  - Local Institution, Sheffield, South Yorkshire
  - Local Institution, Sutton, Surrey
  - Local Institution, Newcastle upon Tyne, Tyne and Wear
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Cambridge

REFERENCES:
- [Derived] Hunger SP, Tran TH, Saha V, Devidas M, Valsecchi MG, Gastier-Foster JM, Cazzaniga G, Reshmi SC, Borowitz MJ, Moorman AV, Heerema NA, Carroll AJ, Martin-Regueira P, Loh ML, Raetz EA, Schultz KR, Slayton WB, Cario G, Schrappe M, Silverman LB, Biondi A. Dasatinib with intensive chemotherapy in de novo paediatric Philadelphia chromosome-positive acute lymphoblastic leukaemia (CA180-372/COG AALL1122): a single-arm, multicentre, phase 2 trial. Lancet Haematol. 2023 Jul;10(7):e510-e520. doi: 10.1016/S2352-3026(23)00088-1. PMID 37407142
- [Derived] Tasian SK, Peters C. Targeted therapy or transplantation for paediatric ABL-class Ph-like acute lymphocytic leukaemia? Lancet Haematol. 2020 Dec;7(12):e858-e859. doi: 10.1016/S2352-3026(20)30369-0. No abstract available. PMID 33242441
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 106 participants were treated with dasatinib.
Groups:
- Dasatinib Cohort: Children and adolescents newly diagnosed with Philadelphia chromosome positive acute lymphocytic leukemia (Ph+ ALL) treated with standard multiagent chemotherapy and Dasatinib (either in tablets or Powder For Oral Suspension (PFOS)) at a dose of 60 mg/m2 daily.
Period: Treatment Phase
Arm/Group | Dasatinib Cohort
Started | 106
Completed | 78
Not Completed | 28
Not completed — Lack of Efficacy | 3
Not completed — Study Drug Toxicity | 2
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 4
Not completed — Death | 2
Not completed — Other reasons | 9
Period: Follow-up Phase
Arm/Group | Dasatinib Cohort
Started | 100 (Some of the participants who did not completed the Treatment Phase were still moved to the Follow-up Phase)
Completed (Completed = continuing in the follow-up phase) | 0
Not Completed | 100
Not completed — Withdrawal by Subject | 4
Not completed — Death | 14
Not completed — Lost to Follow-up | 7
Not completed — Follow-up no longer required per protocol | 70
Not completed — Other and not reported reasons | 5

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib Cohort
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All treated particpants
  Years | 9.29 (4.467)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated particpants
  Participants
    Female | 49
    Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 27
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    American Indian or Alaska Native | 1
    Asian | 5
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 13
    White | 85
    More than one race | 0
    Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: 3-year Event-free Survival (EFS) Rate
Description: 3-year EFS rate is defined as the percentage of participants without event after 3 years since the start of study treatment.
  Events for EFS are defined as ANY first one of the following:
  * Lack of complete response in bone marrow
  * Relapse at any site
  * Development of second malignant neoplasm
  * Death from any cause
Time Frame: From first dose to 3 years following first dose
Population: All treated partcipants
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dasatinib Cohort
Number analyzed (Participants) | 106
Percentage of Participants | 66.0 [57.7 to 73.7]
Statistical Analysis 1: Comparison: Dasatinib Cohort; Difference in 3-year binomial EFS rate in all treated participants (dasatinib plus chemotherapy) vs. chemotherapy alone in AIEOP-BFM 2000 historical control; Test type: Superiority; p = 0.032, Chi-squared — Superiority test versus AIEOP-BFM 2000; Estimate of Difference = 16.86, 90% CI 2-sided [3.9 to 29.8] — Treatment difference (CA180372 - AIEOP-BFM 2000)
Statistical Analysis 2: Comparison: Dasatinib Cohort; Difference in 3-year binomial EFS rate for all treated participants (dasatinib plus chemotherapy) vs. continuous imatinib plus chemotherapy in the Amended EsPhALL Trial Historical Control; Test type: Non-Inferiority — non-inferiority margin = 5%. One-sided type I error rate of 0.05; p = 0.271, Chi-squared — Superiority test versus EsPhALL; Estimate of difference = 6.91, 90% CI 2-sided [-3.3 to 17.2] — Treatment difference (CA180372 - EsPhALL) Test if lower confidence limit is above -5%
Statistical Analysis 3: Comparison: Dasatinib Cohort; Test type: Superiority — Difference in 3-year binomial EFS rate in all treated participants (dasatinib plus chemotherapy) vs. chemotherapy alone in COG AALL0031 historical control; p = 0.157, Chi-squared; Estimate of difference = -10.75, 90% CI 2-sided [-22.7 to 1.2] — Treatment difference (CA180372 - COG AALL0031)

2. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing different types of all causality all grade adverse events
Time Frame: From first dose to 100 days following last dose (up to approximately 23 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib Cohort
Number analyzed (Participants) | 106
Participants
  Adverse Events (AEs) | 106
  Drug-related AEs | 88
  AEs leading to discontinuation | 7
  Serious Adverse Events (SAEs) | 101
  Deaths | 15

3. Secondary Outcome: Event-Free Survival (EFS) Rate (Kaplan-Meier Estimates)
Description: Overall estimation of the EFS of dasatinib plus chemotherapy was performed utilizing the Kaplan-Meier (KM) Product Limit method. The 3-year and 5-year EFS rates were computed with the corresponding 95% CI's using Greenwood's formula. Analyses of EFS included KM plots with number of patients at risk. Participants who neither relapse nor die or who are lost to follow-up were censored on the date of their last bone marrow, CSF assessment or physical exam, whichever occurred last.
Time Frame: From first dose to 3 years or 5 years following first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dasatinib Cohort
Number analyzed (Participants) | 106
Percentage of Participants
  3-year EFS Estimate | 65.5 [55.5 to 73.7]
  5-year EFS Estimate | 53.1 [42.8 to 62.3]

4. Secondary Outcome: Complete Remission Rate
Description: Complete Remission rate is defined as the percentage of participants achieving a complete remission, i.e. < 5% lymphoblasts in bone marrow and in CSF, with no evidence of other extramedullary disease. Complete remission will be assessed at the end of Induction IA, end of induction IB and end of the consolidation period for all treated participants.
Time Frame: From first dose to End of Induction Period Ia (up to 5 weeks) or Ib (up to 9 weeks) or End of Consolidation Period (up to 22 weeks)
Population: All treated participants
Measure: Number; unit: Percentage of Partcipants
Arm/Group | Dasatinib Cohort
Number analyzed (Participants) | 106
Percentage of Partcipants
  End of Induction period Ia | 65.1
  End of Induction period Ib | 88.7
  End of Consolidation period | 93.4

5. Secondary Outcome: Percentage of Participants Negative for Minimal Residual Disease (MRD)
Description: MRD was by real-time qPCR for clone-specific immunoglobulin and T-cell receptor gene rearrangements (IG/TCR). Participants were declared as MRD negative if the MRD level is undetectable providing the assay lower limit of quantification is at least 0.1%
Time Frame: as for outcome 4
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dasatinib Cohort
Number analyzed (Participants) | 106
Percentage of Participants
  End of Induction period Ia | 28.3 [19.98 to 37.88]
  End of Induction period Ib | 52.8 [42.89 to 62.60]
  End of Consolidation period | 71.7 [62.12 to 80.02]

6. Secondary Outcome: Percentage of Participants With BCR-ABL Mutations at Baseline and at Time of Disease Progression or Relapse
Description: A BCR-ABL mutation is defined as the presence of a detectable amino acid substitution in the ABL kinase domain, assessed by Real-time quantitative PCR.
Time Frame: At baseline (prior to start of study treatment) and at disease progression or relapse (up to approximately 3 years)
Population: All treated participants with available measurements
Measure: Number; unit: Percentage of participants
Arm/Group | Dasatinib Cohort
Number analyzed (Participants) | 106
Percentage of participants
  At Baseline: number analyzed (Participants) | 80
  At Baseline | 1.3
  At Disease Progression or Relapse: number analyzed (Participants) | 31
  At Disease Progression or Relapse | 6.5

ADVERSE EVENTS:
Time Frame: All cause mortality was assessed from first dose to study completion. SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 23 months)
Arm/Group | Dasatinib Cohort
All-Cause Mortality (participants affected / at risk) | 21/106
Serious Adverse Events (participants affected / at risk) | 101/106
Other Adverse Events (participants affected / at risk) | 106/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Cohort (N=106)
ANAEMIA (Blood and lymphatic system disorders) | 13
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 81
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 4
LYMPHATIC DISORDER (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 25
PANCYTOPENIA (Blood and lymphatic system disorders) | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 10
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1
SINUS TACHYCARDIA (Cardiac disorders) | 3
TACHYCARDIA (Cardiac disorders) | 2
HYPOACUSIS (Ear and labyrinth disorders) | 1
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1
PHOTOPHOBIA (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 11
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1
ASCITES (Gastrointestinal disorders) | 2
COLITIS (Gastrointestinal disorders) | 10
CONSTIPATION (Gastrointestinal disorders) | 3
DIARRHOEA (Gastrointestinal disorders) | 21
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1
ENTERITIS (Gastrointestinal disorders) | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 2
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1
GASTRIC PERFORATION (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
ILEUS (Gastrointestinal disorders) | 2
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4
NAUSEA (Gastrointestinal disorders) | 6
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 7
OESOPHAGITIS (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1
PROCTALGIA (Gastrointestinal disorders) | 1
PROCTITIS (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 15
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 16
CHILLS (General disorders) | 1
DEVICE RELATED THROMBOSIS (General disorders) | 1
INFLUENZA LIKE ILLNESS (General disorders) | 1
LOCALISED OEDEMA (General disorders) | 1
MUCOSAL INFLAMMATION (General disorders) | 18
NON-CARDIAC CHEST PAIN (General disorders) | 2
OEDEMA (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
PAIN (General disorders) | 3
PYREXIA (General disorders) | 52
CHOLECYSTITIS (Hepatobiliary disorders) | 1
HEPATITIS TOXIC (Hepatobiliary disorders) | 1
VENOOCCLUSIVE LIVER DISEASE (Hepatobiliary disorders) | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 7
DRUG HYPERSENSITIVITY (Immune system disorders) | 7
ABDOMINAL INFECTION (Infections and infestations) | 2
BACTERAEMIA (Infections and infestations) | 14
BACTERIAL SEPSIS (Infections and infestations) | 3
BRONCHITIS (Infections and infestations) | 1
CANDIDA INFECTION (Infections and infestations) | 3
CANDIDA PNEUMONIA (Infections and infestations) | 1
CATHETER SITE INFECTION (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 3
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 6
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 7
COCCIDIOIDOMYCOSIS (Infections and infestations) | 1
CONJUNCTIVITIS (Infections and infestations) | 3
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 14
EMPYEMA (Infections and infestations) | 1
ENTEROCOLITIS BACTERIAL (Infections and infestations) | 2
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 2
ESCHERICHIA SEPSIS (Infections and infestations) | 2
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1
FUNGAL SEPSIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 2
HEPATIC INFECTION (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 3
INFECTION (Infections and infestations) | 2
INFLUENZA (Infections and infestations) | 3
KIDNEY INFECTION (Infections and infestations) | 1
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1
LOCALISED INFECTION (Infections and infestations) | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
LUNG INFECTION (Infections and infestations) | 10
MUCOSAL INFECTION (Infections and infestations) | 2
NAIL BED INFECTION (Infections and infestations) | 1
NAIL INFECTION (Infections and infestations) | 1
NEUTROPENIC INFECTION (Infections and infestations) | 1
OSTEOMYELITIS (Infections and infestations) | 1
OTITIS MEDIA (Infections and infestations) | 5
PASTEURELLA INFECTION (Infections and infestations) | 1
PELVIC INFECTION (Infections and infestations) | 1
PERINEAL CELLULITIS (Infections and infestations) | 1
PERIORBITAL CELLULITIS (Infections and infestations) | 1
PERITONITIS (Infections and infestations) | 2
PHARYNGITIS (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 10
PNEUMONIA BACTERIAL (Infections and infestations) | 1
PNEUMONIA VIRAL (Infections and infestations) | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 1
RASH PUSTULAR (Infections and infestations) | 2
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 20
SEPTIC EMBOLUS (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 6
SINUSITIS (Infections and infestations) | 3
SKIN INFECTION (Infections and infestations) | 4
SPLENIC INFECTION (Infections and infestations) | 1
STREPTOCOCCAL SEPSIS (Infections and infestations) | 1
SYSTEMIC CANDIDA (Infections and infestations) | 1
SYSTEMIC MYCOSIS (Infections and infestations) | 1
TOOTH ABSCESS (Infections and infestations) | 1
TOOTH INFECTION (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 3
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1
VIRAL DIARRHOEA (Infections and infestations) | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1
ANAPHYLACTIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 2
OVERDOSE (Injury, poisoning and procedural complications) | 1
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 2
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3
BLOOD BILIRUBIN INCREASED (Investigations) | 2
BLOOD CREATININE INCREASED (Investigations) | 7
BLOOD CULTURE POSITIVE (Investigations) | 1
DRUG CLEARANCE DECREASED (Investigations) | 2
ENTEROVIRUS TEST POSITIVE (Investigations) | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 9
PLATELET COUNT DECREASED (Investigations) | 7
TRANSAMINASES INCREASED (Investigations) | 1
TROPONIN I INCREASED (Investigations) | 1
URINE OUTPUT DECREASED (Investigations) | 1
VIRAL TEST (Investigations) | 2
WEIGHT DECREASED (Investigations) | 3
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 6
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
DEHYDRATION (Metabolism and nutrition disorders) | 11
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9
HYPONATRAEMIA (Metabolism and nutrition disorders) | 8
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ASTROCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LEUKAEMIA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1
DYSARTHRIA (Nervous system disorders) | 1
ENCEPHALOPATHY (Nervous system disorders) | 2
FACIAL PARESIS (Nervous system disorders) | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 8
HEMIPARESIS (Nervous system disorders) | 1
LEUKOENCEPHALOPATHY (Nervous system disorders) | 2
PARAESTHESIA (Nervous system disorders) | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 4
PRESYNCOPE (Nervous system disorders) | 1
SEIZURE (Nervous system disorders) | 5
ANXIETY (Psychiatric disorders) | 1
DELIRIUM (Psychiatric disorders) | 2
PERSONALITY CHANGE (Psychiatric disorders) | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 10
BLADDER SPASM (Renal and urinary disorders) | 1
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1
OEDEMA GENITAL (Reproductive system and breast disorders) | 1
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 8
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 7
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 9
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 3
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1
EMBOLISM (Vascular disorders) | 3
HYPERTENSION (Vascular disorders) | 7
HYPOTENSION (Vascular disorders) | 22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Cohort (N=106)
ANAEMIA (Blood and lymphatic system disorders) | 83
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 37
LEUKOPENIA (Blood and lymphatic system disorders) | 12
NEUTROPENIA (Blood and lymphatic system disorders) | 43
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 50
PERICARDIAL EFFUSION (Cardiac disorders) | 6
SINUS TACHYCARDIA (Cardiac disorders) | 19
TACHYCARDIA (Cardiac disorders) | 35
EAR PAIN (Ear and labyrinth disorders) | 25
EYE PAIN (Eye disorders) | 8
OCULAR HYPERAEMIA (Eye disorders) | 7
PERIORBITAL OEDEMA (Eye disorders) | 9
VISION BLURRED (Eye disorders) | 15
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 11
ABDOMINAL PAIN (Gastrointestinal disorders) | 73
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 19
ANAL INFLAMMATION (Gastrointestinal disorders) | 7
COLITIS (Gastrointestinal disorders) | 13
CONSTIPATION (Gastrointestinal disorders) | 58
DIARRHOEA (Gastrointestinal disorders) | 75
DYSPEPSIA (Gastrointestinal disorders) | 7
HAEMATOCHEZIA (Gastrointestinal disorders) | 14
MOUTH ULCERATION (Gastrointestinal disorders) | 8
NAUSEA (Gastrointestinal disorders) | 81
ORAL PAIN (Gastrointestinal disorders) | 27
PROCTALGIA (Gastrointestinal disorders) | 15
STOMATITIS (Gastrointestinal disorders) | 49
TOOTHACHE (Gastrointestinal disorders) | 9
VOMITING (Gastrointestinal disorders) | 83
ASTHENIA (General disorders) | 11
CATHETER SITE ERYTHEMA (General disorders) | 6
CATHETER SITE PAIN (General disorders) | 14
CHILLS (General disorders) | 20
FACE OEDEMA (General disorders) | 8
FATIGUE (General disorders) | 58
GAIT DISTURBANCE (General disorders) | 10
INFLUENZA LIKE ILLNESS (General disorders) | 6
MALAISE (General disorders) | 7
MUCOSAL INFLAMMATION (General disorders) | 51
NON-CARDIAC CHEST PAIN (General disorders) | 18
OEDEMA (General disorders) | 10
OEDEMA PERIPHERAL (General disorders) | 17
PAIN (General disorders) | 28
PYREXIA (General disorders) | 79
DRUG HYPERSENSITIVITY (Immune system disorders) | 17
CANDIDA INFECTION (Infections and infestations) | 11
CELLULITIS (Infections and infestations) | 10
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 11
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 8
CONJUNCTIVITIS (Infections and infestations) | 12
DEVICE RELATED INFECTION (Infections and infestations) | 7
EAR INFECTION (Infections and infestations) | 7
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 10
INFLUENZA (Infections and infestations) | 7
LUNG INFECTION (Infections and infestations) | 8
ORAL CANDIDIASIS (Infections and infestations) | 14
OTITIS MEDIA (Infections and infestations) | 11
PHARYNGITIS (Infections and infestations) | 10
PNEUMONIA (Infections and infestations) | 6
RHINITIS (Infections and infestations) | 11
RHINOVIRUS INFECTION (Infections and infestations) | 7
SEPSIS (Infections and infestations) | 7
SINUSITIS (Infections and infestations) | 18
SKIN INFECTION (Infections and infestations) | 12
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 39
URINARY TRACT INFECTION (Infections and infestations) | 14
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 13
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 6
CONTUSION (Injury, poisoning and procedural complications) | 32
SKIN ABRASION (Injury, poisoning and procedural complications) | 8
SUNBURN (Injury, poisoning and procedural complications) | 7
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 6
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 42
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 35
BLOOD BILIRUBIN INCREASED (Investigations) | 12
BLOOD CREATININE INCREASED (Investigations) | 9
CARDIAC MURMUR (Investigations) | 12
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 6
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 7
LYMPHOCYTE COUNT DECREASED (Investigations) | 8
NEUTROPHIL COUNT DECREASED (Investigations) | 41
PLATELET COUNT DECREASED (Investigations) | 39
WEIGHT DECREASED (Investigations) | 26
WEIGHT INCREASED (Investigations) | 11
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 21
DECREASED APPETITE (Metabolism and nutrition disorders) | 40
DEHYDRATION (Metabolism and nutrition disorders) | 14
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 23
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 34
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 30
HYPOKALAEMIA (Metabolism and nutrition disorders) | 50
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 19
HYPONATRAEMIA (Metabolism and nutrition disorders) | 23
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 23
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 38
BACK PAIN (Musculoskeletal and connective tissue disorders) | 48
BONE PAIN (Musculoskeletal and connective tissue disorders) | 22
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 21
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 8
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 15
MYALGIA (Musculoskeletal and connective tissue disorders) | 15
NECK PAIN (Musculoskeletal and connective tissue disorders) | 9
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 63
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 18
DIZZINESS (Nervous system disorders) | 14
HEADACHE (Nervous system disorders) | 70
LETHARGY (Nervous system disorders) | 7
NEUROPATHY PERIPHERAL (Nervous system disorders) | 6
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 12
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 13
TREMOR (Nervous system disorders) | 8
AGITATION (Psychiatric disorders) | 10
ANXIETY (Psychiatric disorders) | 15
DEPRESSION (Psychiatric disorders) | 16
INSOMNIA (Psychiatric disorders) | 16
IRRITABILITY (Psychiatric disorders) | 12
DYSURIA (Renal and urinary disorders) | 12
HAEMATURIA (Renal and urinary disorders) | 13
URINARY RETENTION (Renal and urinary disorders) | 6
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 8
COUGH (Respiratory, thoracic and mediastinal disorders) | 78
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 18
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 27
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 15
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 28
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 35
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 16
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 8
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 10
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 8
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 37
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 7
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 11
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 13
ALOPECIA (Skin and subcutaneous tissue disorders) | 21
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 9
DRY SKIN (Skin and subcutaneous tissue disorders) | 19
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 7
ERYTHEMA (Skin and subcutaneous tissue disorders) | 22
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 6
PETECHIAE (Skin and subcutaneous tissue disorders) | 17
PRURITUS (Skin and subcutaneous tissue disorders) | 27
RASH (Skin and subcutaneous tissue disorders) | 48
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 21
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 8
SWELLING FACE (Skin and subcutaneous tissue disorders) | 9
URTICARIA (Skin and subcutaneous tissue disorders) | 9
FLUSHING (Vascular disorders) | 10
HAEMATOMA (Vascular disorders) | 6
HYPERTENSION (Vascular disorders) | 41
HYPOTENSION (Vascular disorders) | 28
PALLOR (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2013-10-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT01460160/Prot_000.pdf
  • Statistical Analysis Plan (2013-10-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT01460160/SAP_001.pdf